CLINICAL TRIAL: NCT01428726
Title: A Phase IIa Multicenter Double Blind Study to Evaluate the Efficacy and Safety of Low Doses of Oral NT-KO-003 for the Treatment of Multiple Sclerosis
Brief Title: A Phase IIa Study of NT-KO-003 for Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotec Pharma (Industry)
Collaborators: Advancell - Advanced In Vitro Cell Technologies, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT-KO-003-2010-01
Record Dates: First submitted 2011-08-31; First posted 2011-09-05 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: NT-KO-003; RRMS; efficacy; safety; Phase IIa
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: NT-KO-003
- NT-KO-003 low dose (Experimental)
  Interventions: Drug: NT-KO-003
- NT-KO-003 high dose (Experimental)
  Interventions: Drug: NT-KO-003

INTERVENTIONS:
Drug: NT-KO-003 — NT-KO-003 is a coated tablet, administered once a day

SUMMARY:
The aim of the study is to assess the efficacy and safety of NT-KO-003 in the treatment of relapsing remitting multiple sclerosis, comparing two doses versus placebo.

DETAILED DESCRIPTION:
This is a Phase IIa study, double blind, placebo Controlled, Multicenter Study that will involve up to 99 patients with relapsing remitting multiple sclerosis.

After signing the informed consent form, subjects will be randomized to three treatments arms: placebo, NT-KO-003 low dose or NT-KO-003 high dose. Treatment will continue daily during 6 months. A MRI and a clinical evaluation will be performed monthly. Safety will be assessed during the 6 months treatment and until 15 days after the finalization of the treatment.

Patients will be allowed to continue in the same arm of the study, in a blinded way, until the study finalizes as optional extension treatment. Patient will sign the Extension Informed Consent and a MRI will be performed for those patients still in treatment after 12 months of the inclusion in the core study (visit 0).

ELIGIBILITY:
Inclusion Criteria

* Patients who meet the diagnosis criteria for MS according to guidelines provided by McDonald et al (1)
* Patients who meet the diagnosis criteria for RRMS
* Patients with clinical disability measured by EDSS score between 0 and 5.0 inclusive
* Patients who present at least 1 relapse in the previous 2 years or presence of at least 1 gadolinium-enhanced lesion in the previous 1 year
* Patients aged between 18 to 55 years old, either gender

Exclusion Criteria

* Patients who are candidates for treatment with drugs modifying the course of the disease according to the criteria of the Regulatory Agencies in each country, unless the patient refuses to initiate such therapy or decide to postpone the start of this therapy
* Patients with relapse in the 30 days period before baseline visit
* Patients in treatment with NT-KO-003
* Medical conditions such as hypotension, insulinoma, hyperuricemia
* Patients with Diabetes defined by ADA criteria (2)
* Other conditions: drug abuse, inability to consent, or inability to perform all the procedures for the Clinical Trial
* Contraindications for MRI studies: claustrophobia, heart pacemaker or any other condition that would preclude proximity to strong magnetic field
* Contraindications for treatment with NT-KO-003 or excipients: allergies, hypersensitivity
* Patients with known allergy or with contraindications to the administration of intravenous gadolinium-based agents (chronic or acute renal failure according to The Renal Association or NICE guidelines (3))
* Corticosteroid therapy in the last month
* Interferon-beta or Glatiramer acetate therapy in the last 3 months
* Natalizumab therapy in the last 6 months
* Patients treated with chemotherapy (Mitoxantrone, Azathioprine, Cyclophosphamide, Cladribine, Methotrexate) or monoclonal antibodies that deplete populations of cells (rituximab, alemtuzumab, ocrelizumab, daclizumab) in the last 12 months or have entered in previous trials with treatments in development in the last 3 months
* Patients participating in another Clinical Trial at the moment of the screening visit
* Patient who had received a liver transplantation or candidates for liver transplantation
* Positive pregnancy test, breast feeding women or of childbearing potential not using highly effective methods of contraception
* Male patients that do not follow adequate contraceptive measurements
* Fingolimod therapy in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of NT-KO-003 in patients with relapsing remitting MS patients | 6 months
  efficacy will be measured as the cumulative number of new lesions observed in all MRIs, with exception of baseline

SECONDARY OUTCOMES:
Efficacy of NT-KO-003 in relapsing remitting MS patients | 6 months
  efficacy measured as the cumulative number of new lesions (gadolinium enhanced lesions and T2 lesions) in all MRIs
Clinical efficacy of NT-KO-003 in relapsing remitting MS patients | 6 months
  clinical efficacy will be measured as relapse rates and EDSS scale
Safety of NT-KO-003 in patients with relapsing remitting MS patients | six and a half months
  safety will be measured as the incidence of adverse events and serious adverse events (incidence, causality, and severity) related to treatment with NT-KO-003

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Villoslada, MD PhD, Principal Investigator — Hospital Clinic i Provincial de Barcelona, Spain
Locations (17):
- Germany (3):
  - Charité Universitätsmedizin, Berlin
  - Klinik und Poliklinik für Neurologie, Münster
  - Neurologisches Studienzentrum an der Stiftung Deutsche Klinik für Diagnostik GmbH, Wiesbaden
- Spain (14):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Universitari Josep Trueta, Girona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Puerta del Hierro, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario La Fe, Valencia
  - Hospital Xeral Vigo, Vigo